CLINICAL TRIAL: NCT03181243
Title: The Acceptance, Safety, and Efficacy of Needle-free Jet Anaesthetic Technique (MadaJet) Versus Needle Injection for Sperm Retrieval in Patients With Azoospermia
Brief Title: The Acceptance, Safety, and Efficacy of MadaJet Versus Needle Injection for Sperm Retrieval in Patients With Azoospermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam National University (Other)
Responsible Party: Principal Investigator, Manh Tuong Ho, Director, Vietnam National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCKH/CGRH_03_2017
Record Dates: First submitted 2017-06-02; First posted 2017-06-08 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male | interventions — Needles

STUDY DESIGN:
Intervention Model Description: Because the length of sperm retrieval procedure is significantly different between groups, we use matched pairs based on the length of procedure as the matching variable for the primary outcome (pain relief) by specify two in one block. We create a block 2 to assign sample numbers equally to each group (MadaJet or needle injection) and assign equitably the block to each procedure (TESE or PESA). Therefore, patients will be randomized, using a computer-generated randomization list in a 1:1 ratio and block 2, to either the MadaJet group or to needle injection group after the assessment of eligibility and signing informed consents. Allocation of patients will be done by a third-party via telephone according to the specified list. The patients don't know which anaesthesia technique will be performed.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MadaJet (Experimental): Jet injector (Madajet medical Urology) preloaded as manufacturer's instruction
  Interventions: Procedure: Madajet
- Needle injection (Experimental): 01 sterile 10-mL syringe with small gauge needle (25 ga), solution for sterile preparation, 10 - 15 mL Lidocaine 2%
  Interventions: Procedure: Needle injection

INTERVENTIONS:
Procedure: Madajet — The spermatic cord is firmly trapped between the middle finger, index finger and thumb of the left hand. The injector's sheath is placed over the spermatic cord with gentle pressure adjacent to the external inguinal ring. Depending upon the thickness of spermatic cord, three or four injections are consecutively administered around it, beginning from proximal to distal points.
  Other Names: Needle-free jet anaesthetic technique
  Arms: MadaJet
Procedure: Needle injection — The pubic tubercle is palpated on the side that is going to be blocked. The spermatic cord is then immobilised with the non-dominant hand between the thumb and index finger. Right after needle puncture with attached syringe and local anaesthetic solution is conducted at a point that is 1 cm inferior to and 1 cm medial to the pubic tubercle, pass the needle directly downward in a vertical fashion, which leads it into the spermatic cord. After a check-up (negative aspiration) for bleeding, approximately 3 mL of solution (Lidocaine 2%) is injected into the cord.
  Other Names: Local aesthesia by needle injection
  Arms: Needle injection

SUMMARY:
To compare the acceptance, safety, and efficacy of needle-free jet anaesthetic technique (MadaJet) versus needle injection for sperm retrieval in patients with azoospermia.

DETAILED DESCRIPTION:
Azoospermia is found in 1-3% of general population and 10-15% of men presenting with infertility. In this scenario, there are no spermatozoa in the patient's semen after centrifugation, and pregnancy may be achieved through IVF/ Intracytoplasmic sperm injection (ICSI) combined with sperm retrieval techniques (e.g. PESA, testicular sperm extraction - TESE, TESA). These techniques are commonly conducted under local anesthesia, which a 10-15 mL solution of 2% lidocaine hydrochloride injected around the spermatic cord near the external inguinal ring. However, needle fear is prevalent in both children (~33-63%) and adults (~14-38%) and can contribute to negative experiences with needle procedures and health care for patients, caregivers, and health professionals. In clinical practice, patients often concern about the pain, trauma and possible complication (i.e. wheal, hematoma, infection) of needle injection of local anaesthesia into and through the scrotal wall when performing sperm retrieval. It not only interferes with clinicians' abilities to carry out procedures (e.g. due to flailing and attempts to escape), but also undermines the efficacy of pain interventions at the time of the needle. Therefore, receiving local anaesthesia without a needle is easily well accepted by the patients with azoospermia.

The needleless jet injector (MadaJet Medical Injector) has been widely used in the fields of dermatology, cosmetic and plastic surgery, gynecology, dentistry, and podiatry as well as for immunization. It was also employed for no-scalpel vasectomy in Urology/Andrology. The first studies using needleless jet injector for spermatic cord block was reported by Wilson in 2001 and Weiss in 2005. The next studies showed that MadaJet has better outcomes (e.g. cost, pain scores, onset time) than traditional needle anaesthesia (16-18). Unlike a conventional spermatic cord block with needle injection, there is no wheal on the patients' skin and local edema after administering injection. A mist of solution with a high-pressure injector will be rapidly delivered and absorbed through the skin to the tissue beneath around the cord with much less trauma. As a consequence, it is less painful than the needle injection.

For those reasons, a needle-free jet anaesthetic technique for sperm retrieval will be described for local anaesthesia, which may minimize the fear of the needle. The acceptance, safety, and efficacy of this technique will also be compared with needle injection for sperm retrieval in azoospermia patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients (including obstructive azoospermia and non-obstructive azoospermia) in need of sperm retrieval (PESA, TESE) for ICSI.

Exclusion Criteria:

* Have not finished the process of sperm retrieval techniques.
* Malformation of genital organs (e.g. spermatic cord, testicle)
* Anxious, alcoholic patients.
* Patients giving a history of personality disorders.
* Patients who abuse drugs.
* Disagree to participate in the study.

Ages: 20 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2017-12-25 (Actual); Study Completion 2017-12-25 (Actual)

PRIMARY OUTCOMES:
Pain score | 1 year
  Right after completing the injection, information about the pain before, during and after the sperm retrieval technique will be immediately documented by the visual analog scale (VAS) questionnaire on 10 cm lines (0 represents no pain, whereas 10 marks the highest score).

SECONDARY OUTCOMES:
Pressure (fear) of the patients | 1 year
  Right after completing the injection, information about the pain before, during and after the sperm retrieval technique will be immediately documented by the visual analog scale (VAS) questionnaire on 10 cm lines (0 represents no pain, whereas 10 marks the highest score).
Discomfort of the patients | 1 year
  Right after completing the injection, information about the pain before, during and after the sperm retrieval technique will be immediately documented by the visual analog scale (VAS) questionnaire on 10 cm lines (0 represents no pain, whereas 10 marks the highest score).
Incidence of treatment (Bleeding) | 1 year
  Bleeding will be recorded peri- and post- operative anesthesia.
Incidence of treatment (Swelling) | 1 year
  Swelling will be recorded peri- and post- operative anesthesia.
Incidence of treatment (Hematoma) | 1 year
  Hematoma will be recorded peri- and post- operative anesthesia.
Onset of action of Madajet | 1 year
  By using the stopwatch, the onset of action of anesthesia will be recorded. Every five seconds, the pain reaction which shows the onset is determined on the scrotum by using tissue forceps.
Duration of action of Madajet | 1 year
  By using the stopwatch, the duration of action of anesthesia will be recorded. The patients are observed in the operation room until all the symptoms of anesthesia wore off. The total duration of anesthesia is measured from the time of onset until the patient reports normal reaction in the scrotum.
Onset of action of Needle injection | 1 year
  By using the stopwatch, the onset of action of anesthesia will be recorded. Every thirty seconds, the pain reaction which shows the onset is determined on the scrotum by using tissue forceps.
Duration of action of Needle injection | 1 year
  By using the stopwatch, the duration of action of anesthesia will be recorded. The patients are observed in the operation room until all the symptoms of anesthesia wore off. The total duration of anesthesia is measured from the time of onset until the patient reports normal reaction in the scrotum.

CONTACTS AND LOCATIONS:
Overall Officials: Khoa D Le, Dr, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No